CLINICAL TRIAL: NCT02515409
Title: Heated Humidified High Flow Nasal Cannula for Children With Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-15-KA-0263-15-TLV-CTIL
Record Dates: First submitted 2015-06-28; First posted 2015-08-04 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-06

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea Syndrome (OSAS); Heated Humidified High Flow Nasal Cannula (HHHNC); Continues positive airway pressure (CPAP); Children; Non invasive ventilation; Treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CPAP: CPAP, as a first line treatment to OSAS.
  Interventions: Device: CPAP
- HHHFNC: Treatment with HHHFNC after CPAP treatment fails.
  Interventions: Device: HHHFNC

INTERVENTIONS:
Device: HHHFNC — After the treatment with CPAP fails, the participants will use HHHFNC as a treatment for OSAS.
  Groups: HHHFNC
Device: CPAP — CPAP, as a first line treatment in OSAS.
  Groups: CPAP

SUMMARY:
The purpose of this study is to determine whether heated humidified high flow nasal cannula (HHHFNC) is effective as a treatment of obstructive sleep apnea syndrome (OSAS) compared to continues positive airway pressure (CPAP) treatments in children and to compare their adherence and compliance.

ELIGIBILITY:
Inclusion criterias:

* Age: 0-16 years old.
* Refered for treatment with non invasive ventilation.
* Diagnosed with OSAS and AHI>=5

There are no exclusion criteria

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children ages 0-16 years with obstractive sleep apnea, referred for treatment with non invasive ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Average hours per night and per week using HHHFNC . | One year
Average hours per night and per week using CPAP. | One year

SECONDARY OUTCOMES:
Apnea hypopnea index (AHI) | One year
  Severity of sleep apnea using AHI.
Pediatric sleep questionnaire (PSQ) score | One year
  Obstructive sleep-related breathing disorders using PSQ score

CONTACTS AND LOCATIONS:
Overall Officials: Keren Armoni-Domany, Dr., Principal Investigator — Tel-Aviv Sourasky Medical Center